CLINICAL TRIAL: NCT03929874
Title: Ultrasound Image Study for Ultrasound-assisted Paramedian Spinal Anesthesia: Difference in Sidedness of Approach, Position and Age
Brief Title: Ultrasound Image Study for Ultrasound-assisted Paramedian Spinal Anesthesia
Status: Completed | Type: Observational
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Jin-Tae Kim, Professor, Seoul National University Hospital
Other Study IDs: H-1903-110-1018
Record Dates: First submitted 2019-04-25; First posted 2019-04-29 (Actual); Last update posted 2019-07-11 (Actual); Status verified 2019-07

CONDITIONS: Anesthesia, Spinal; Ultrasonography; Sidedness; Position

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- 18 ≤ age ≤ 40: 18 ≤ age ≤ 40
- age ≥ 60: age ≥ 60

SUMMARY:
This prospective observational study aimed to obtain ultrasound images for ultrasound-assisted paramedian spinal anesthesia and identify the differences according to sidedness of approach, position and age.

ELIGIBILITY:
Inclusion Criteria:

* Patients under 40 or over 60 years of age who require spinal anesthesia for orthopedic surgery,
* with ASA physical status classification system I, II, III

Exclusion Criteria:

* Patients with contraindication to spinal anesthesia (coagulopathy, local infection, allergy to local anesthetic)
* Patients with communication difficulties
* Patient who can not take a sitting or lateral decubitus position (fracture)
* Patients with a history of spinal surgery
* Patient with anatomical abnormality of the spine

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients under 40 orover 60 years of age who require spinal anesthesia for orthopedic surgery, with ASA physical status classification system I, II, III
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2019-05-02 (Actual); Primary Completion 2019-06-19 (Actual); Study Completion 2019-06-30 (Actual)

PRIMARY OUTCOMES:
Ultrasonic visualization grading at left L3-4, L4-5, L5-S1 interspace and right L3-4, L4-5, L5-S1 interspace in lateral decubitus position and sitting position | Preanesthesia
  * Good: Both LFD (ligamentum flavum-dura mater complex) and PLL (posterior longitudinal ligament) are visible
  * Intermediate: Only one of LFD or PLL is visible
  * Poor: LFD and PLL are not visible
Distance between the midline and the expected location of needle insertion | Preanesthesia
  Distance between the midline of the vertebrae and the expected location of needle insertion at left L3-4, L4-5, L5-S1 interspace and right L3-4, L4-5, L5-S1 interspace in lateral decubitus position and sitting position
Height of LFD through interlaminar space | Preanesthesia
  Height of LFD through interlaminar space visible in ultrasound image at left L3-4, L4-5, L5-S1 interspace and right L3-4, L4-5, L5-S1 interspace in lateral decubitus position and sitting position
Depth from skin to LFD | Preanesthesia
  The depth from skin to LFD at left L3-4, L4-5, L5-S1 interspace and right L3-4, L4-5, L5-S1 interspace in lateral decubitus position and sitting position
Depth from skin to PLL | Preanesthesia
  The depth from skin to PLL at left L3-4, L4-5, L5-S1 interspace and right L3-4, L4-5, L5-S1 interspace in lateral decubitus position and sitting position
Width of the intrathecal space | Preanesthesia
  The distance between the LFD and the PLL at left L3-4, L4-5, L5-S1 interspace and right L3-4, L4-5, L5-S1 interspace in lateral decubitus position and sitting position

CONTACTS AND LOCATIONS:
Overall Officials: Jin-Tae Kim Kim, MD, PhD, Principal Investigator — Seoul National University Hospital
Locations (1):
- Seoul national university hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Chin KJ, Perlas A, Chan V, Brown-Shreves D, Koshkin A, Vaishnav V. Ultrasound imaging facilitates spinal anesthesia in adults with difficult surface anatomic landmarks. Anesthesiology. 2011 Jul;115(1):94-101. doi: 10.1097/ALN.0b013e31821a8ad4. PMID 21572316
- [Derived] Bae J, Park SK, Yoo S, Lim YJ, Kim JT. Influence of age, laterality, patient position, and spinal level on the interlamina space for spinal puncture. Reg Anesth Pain Med. 2019 Nov 4:rapm-2019-100980. doi: 10.1136/rapm-2019-100980. Online ahead of print. PMID 31690644